CLINICAL TRIAL: NCT03860454
Title: The Deep Phenotype of Lamin A/C Cardiomyopathy - A Proof-of-principle Relax-omic Pipeline
Brief Title: The Deep Phenotype of Lamin A/C Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Barts Cardiovascular registry (Unknown)
Responsible Party: Sponsor
Other Study IDs: 16/0661; 17/LO/0167 (Other: REC reference)
Record Dates: First submitted 2019-01-15; First posted 2019-03-04 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Lamin A/C Gene Mutation; Dilated Cardiomyopathy, Familial
Keywords: Dilated Cardiomyopathy; Lamin A/C Cardiomyopathy; Heart failure
MeSH Terms: conditions — familial dilated cardiomyopathy; Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lamin DCM (LMNA+): Adults with known pathogenic lamin (LMNA+) gene mutation.
- Wild types DCM (DCMwt): Adults with heart muscle failure but normal (wild-type) LMNA gene (DCMwt).
- Healthy Volunteers (HV): Matched healthy volunteers (HV).

SUMMARY:
This study seeks to discover clinically useful tests to improve the diagnosis of a rare and serious heart muscle disease caused by mutations in a gene called 'Lamin'.

Patients born with lamin gene mutations have apparently healthy hearts initially, they begin experiencing symptoms in their twenties or thirties, and by age 45 the majority have undergone a heart transplant, experienced a major cardiac complication, or have died. Sudden heart rhythm abnormalities are a major cause of sudden death so earlier diagnosis can save lives by enabling timely treatment or implantation of specialised pacemakers (defibrillators). In clinical practice, diagnosis of lamin heart disease currently relies on the genetic test. Very little is known about the detailed imaging features of the hearts of patients with lamin heart disease although advanced echocardiography and cardiac MRI now offer the opportunity to study the health of the heart without the need for radiation.

DETAILED DESCRIPTION:
* Research participants will undergo resting 12-lead ECG, 24-hour ambulatory ECG, baseline echocardiography, exercise echocardiography, cardiac MRI scan.
* Blood samples will be collected in all participants from both centers for immediate laboratory testing.
* Blood and urine samples will be collected in all participants and used for metabolomic, proteomic and lipidomic profiling and for targeted metabolite and enzyme analysis.
* Blood samples will be collected in all participants for future gene code analysis (DNA / RNA).

ELIGIBILITY:
Inclusion Criteria:

* LMNA+ cases with pathogenic LMNA mutations for LMNA+ and heart myocardial samples from the explanted hearts of LMNA+ patients who are scheduled to undergo clinically indicated heart transplantation at the Papworth Hospital NHS Trust.
* DCMWT cases: patients with heart muscle failure but with wild-type lamin gene. Heart myocardial samples from the explanted hearts of DCMWT patients who are scheduled to undergo clinically indicated heart transplantation at the Papworth Hospital NHS Trust.
* HV (controls): matched to cases.

Exclusion Criteria:

* Needle-phobia that would preclude blood-letting
* Participants unwilling to consent
* Patients that have a conventional contraindication for cardiac magnetic resonance imaging (MRI).
* Patients that have had a blood transfusion within the last month and patients having haemodialysis will be excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults with known pathogenic lamin (LMNA+) gene mutations, adults with heart muscle failure but normal (wild-type) LMNA gene (DCMWT) and matched healthy volunteers (HV).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-03-07 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Positive and negative predictive value of imaging-omics test for diagnosing LMNA-related heart muscle disease. | 3-4 years

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - University Hospital Birmingham (UHB), Birmingham
  - Barts Heart Center, St Bartholomew's Hospital NHS Trust, London
  - Royal Brompton Hospital NHS Trust (RBHT), London
  - Royal Free Hospital NHS Trust (RFH), London
  - University College London Hospital NHS Trust (UCLH), London
  - Papworth Hopsital NHS Trust, Papworth Everard

IPD SHARING:
Plan to Share IPD: No
no sharing of individual patient data is planned.

REFERENCES:
- [Derived] Topriceanu CC, Al-Farih M, Joy G, Chan F, Webber M, Ilie-Ablachim DC, Shiwani H, Tamang M, Banks C, Pettit S, Petersen SE, O'Brien B, Hughes AD, Pierce I, Moody WE, Steeds RP, Puddu PE, Kellman P, Savvatis K, Mohiddin S, Moon JC, Barison A, Piras P, Captur G. The Cardiovascular Magnetic Resonance Phenotype of Lamin Heart Disease. JACC Cardiovasc Imaging. 2025 Jun;18(6):644-660. doi: 10.1016/j.jcmg.2025.01.004. Epub 2025 May 14. PMID 40372342